CLINICAL TRIAL: NCT01816633
Title: A Multi-Center, Prospective, Cohort Trial Comparing the Effectiveness of AutoloGel Therapy to Usual and Customary Care in All Wagner Grades of Diabetic Foot Ulcers
Brief Title: Effectiveness of AutoloGel Therapy in Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol study design was re-done in collaboration with CMS
Sponsor: Cytomedix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM002
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Diabetic Foot Ulcers
Keywords: non healing wound
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AutoloGel (Experimental): Subjects will be treated on average twice a week for the first 2 weeks, and then, once a week thereafter while under active treatment, but actual frequency of treatment will be determined by the treating physician. All subjects will receive AutoloGel treatment.
  Interventions: Device: AutoloGel

INTERVENTIONS:
Device: AutoloGel — AutoloGel is a platelet-rich plasma (PRP) gel used in the treatment of non-healing chronic wounds. It will be administered twice weekly for 2 weeks then weekly

SUMMARY:
The aim of this trial is to demonstrate the effectiveness of complete wound healing in a prospective, open-label, case-matched cohort trial in which diabetic foot ulcers (DFU) will be treated using AutoloGel and case-matched against a concurrent cohort of patients receiving undefined Usual and Customary Care (UCC) as provided in up to 30 U.S. Wound Registry Research Network (USWRRN) centers.

DETAILED DESCRIPTION:
AutoloGel is a platelet-rich plasma gel used in the treatment of non-healing chronic wounds. Prospective observational studies of the effectiveness of AutoloGel have demonstrated promising results in regard to the healing of DFUs, including severe Wagner grade 3 and 4 ulcers. The aim of this trial is to demonstrate the effectiveness of complete wound healing in a prospective, open-label, case-matched cohort trial in which diabetic foot ulcers will be treated using AutoloGel to determine the time to heal at 12 weeks. Comparison will be made with a case-matched concurrent cohort of patients receiving undefined Usual and Customary Care (UCC).

ELIGIBILITY:
Inclusion Criteria:

1. Medicare/Medicaid eligible
2. ≥18 years of age
3. Type I or II diabetes requiring medical treatment as determined by the physician
4. The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (Index Ulcer) is a Wagner 1-5 DFU (see Appendix 9 for Wagner Classification) that is located on the dorsal, plantar, medial, or lateral aspect of the foot or heel (including all toe surfaces)
5. For subjects with potentially multiple eligible DFUs, the largest ulcer will be selected There must be at least 4 cm between the Index Ulcer and other ulcers; if all ulcers are closer than 4 cm, the subject should not be enrolled (screen failure)
6. Debrided ulcer size between 0.5 cm2 and 50 cm2
7. Demonstrated adequate offloading regimen
8. Duration ≥ 1 month at first visit
9. Subject must be willing to comply with the Protocol, which will be assessed by enrolling clinician.

Exclusion Criteria:

1. Subjects known to be sensitive to AutoloGel components (calcium chloride, thrombin, ascorbic acid) and/or materials of bovine origin
2. Presence of another wound that is concurrently treated and might interfere with treatment of the index wound by AutoloGel (malignancy in nearby wound)
3. Ulcer not of DFU pathophysiology (e.g., venous, vasculitic, radiation, rheumatoid, collagen vascular disease, pressure, or arterial etiology)
4. Any malignancy other than non-melanoma skin cancer
5. Subjects who are cognitively impaired and do not have a healthcare proxy
6. Serum albumin of less than 2.5 g/dL
7. Plasma Platelet count of less than 100 x 109/L
8. Hemoglobin of less than 10.5 g/dL
9. Subject has inadequate venous access for repeated blood draw required for AutoloGel Administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Time to heal | 12 weeks
  The primary objective of the trial is to determine the time to heal diabetic foot ulcers treated with Autologel and Standard of Care at 12 weeks DFUs. Comparison will be made with a concurrent cohort of case matched subjects

SECONDARY OUTCOMES:
Ulcer recurrence | 1 year
  Frequency of ulcer recurrence defined as any new ulcer appearing after the index ulcer healed
Incidence of amputations | 1 year
  Frequency of lower extremity amputations; major/minor amputations will be tabulated but not tested.
Proportion of completely healed ulcers | 12 weeks
  Proportion of patients with completely healed diabetic foot ulcers
W-QOL (Quality of life with Chronic Wounds) score | 12 weeks
  Change in mean W-QOL (Quality of life with Chronic Wounds) score between baseline and 12 weeks
Number of patients with adverse events as a measure of tolerability | 12 weeks
  Frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arcadia, California
  - HyperBarxs at Northside Forsyth, Cumming, Georgia